CLINICAL TRIAL: NCT00392899
Title: Randomized Phase III Trial of Adjuvant Chemotherapy With UFT vs. Observation in Curatively Resected Stage II Colon Cancer
Brief Title: Tegafur-Uracil or Observation in Treating Patients With Stage II Colorectal Cancer That Has Been Completely Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Tokyo Medical and Dental University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000512573; TMDU-BRI-CC-05-01
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage II rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Chemotherapy, Adjuvant; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UFT adjuvant therapy group (Active Comparator): UFT is given at a dose of 500-600 mg/day as tegafur in 2 divided doses after meals for 5 days, followed by a 2-day rest. This one-week cycle is repeated for one year. During protocol treatment, clinical findings and laboratory values are evaluated every month. After the completion of protocol treatment, patients are followed-up, according to the schedule defined in the study protocol, for 5 years until recurrence, other malignancy or death is confirmed.
  Interventions: Drug: UFT adjuvant chemotherapy
- Observation group (No Intervention): Patients are followed-up without adjuvant treatment, according to the schedule defined in the study protocol, for 5 years until recurrence, other malignancy or death is confirmed.

INTERVENTIONS:
Drug: UFT adjuvant chemotherapy — UFT is given at a dose of 500-600 mg/day as tegafur in 2 divided doses after meals for 5 days, followed by a 2-day rest. This one-week cycle is repeated for one year.
  Other Names: Adjuvant chemotherapy with tegafur-uracil
  Arms: UFT adjuvant therapy group

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as tegafur-uracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery. Sometimes, after surgery, the tumor may not need more treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether chemotherapy is more effective than observation in treating colorectal cancer.

PURPOSE: This randomized phase III trial is studying tegafur and uracil to see how well they work compared to observation in treating patients with stage II colorectal cancer that has been completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of adjuvant tegafur-uracil vs observation only in patients with curatively resected stage II colorectal cancer.

Secondary

* Compare relapse-free and overall survival of patients treated with these regimens.
* Compare the occurrence of adverse events in patients treated with these regimens.

OUTLINE: This is a randomized, controlled study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo observation.
* Arm II: Patients receive oral tegafur-uracil on days 1-5. Treatment repeats every 7 days for 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 2,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectosigmoid

  * Stage II disease
* Has undergone curative (R0) resection within the past 8 weeks
* No suspicion of hereditary colorectal cancer
* No severe postoperative complications

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC 3,500-12,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 100 IU/L
* Creatinine ≤ 1.5 mg/dL
* Not pregnant or nursing
* Able to take oral medications
* Major organ functions are preserved
* No other active malignancy
* None of the following conditions:

  * Uncontrolled diabetes mellitus
  * Uncontrolled hypertension
  * Myocardial infarction or unstable angina pectoris within the past 6 months
  * Liver cirrhosis
  * Interstitial pneumonia
  * Pulmonary fibrosis
  * Severe emphysema
* No psychiatric disease or other condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy
* No prior or concurrent radiotherapy
* No concurrent prophylactic growth factors
* No concurrent biologic response modifiers

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2025 (Actual)
Dates: Start 2006-10; Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 9 years
  Disease-free survival is defined as the time from date of enrollement until date of recurrence, other malignancies or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall survival | 9 years
  Overall survival is defined as time from date of enrollment until date of death from any cause.
Types and severities of adverse events | 15 months
  Types and severities of adverse events from date of starting protocol treatment until 30 days after date of finishing the treatment are evaluated according to Japanese version of the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) by Translational Research Informatics Center.

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Sugihara, MD, PhD, Study Chair — Tokyo Medical and Dental University
Locations (272):
- Japan (272):
  - Aichi Medical University, Aichi-gun, Aichi-ken
  - Japanese Red Cross Nagoya First Hospital, Nagoya, Aichi-ken
  - Nagoya Central Hospital, Nagoya, Aichi-ken
  - Nagoya Ekisaikai Hospital, Nagoya, Aichi-ken
  - Ban Buntane Houtokukai Hospital, Nagoya, Aichi-ken
  - West Medical Center Jouhoku Municipal Hospital, Nagoya, Aichi-ken
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Nagoya University School of Medicine, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Nagoya Midori Municipal Hospital, Nagoya, Aichi-ken
  - Aichi Cancer Center at Aichi Hospital, Okazaki, Aichi-ken
  - National Hospital Organization Toyohashi Medical Center, Toyohashi, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Koseiren Kamo Hospital, Toyota, Aichi-ken
  - Akita Kumiai General Hospital, Akita, Akita
  - Yamamoto Kumiai General Hospital, Noshiro, Akita
  - Hiraka General Hospital, Yokote, Akita
  - Aomori City Hospital, Aomori, Aomori
  - Asahi General Hospital, Asahi-machi, Chiba
  - Chiba Cancer Center, Chiba, Chiba
  - Chiba University, Chiba, Chiba
  - Teikyo University Chiba Medical Center, Ichihara, Chiba
  - Juntendo Urayasu Hospital, Urayasu-shi, Chiba
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Sumitomo Besshi Hospital, Niihama, Ehime
  - Fukuiken Saiseikai Hospital, Fukui-shi, Fukui
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - National Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kitakyushu Municipal Medical Center, Kitakyushu, Fukuoka
  - University of Occupational and Environmental Health, Kitakyushu-shi, Fukuoka
  - Kurume University School of Medicine, Kurume, Fukuoka
  - Saint Mary's Hospital, Kurume, Fukuoka
  - Social Insurance Tagawa Hospital, Tagawa, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gifu Municipal Hospital, Gifu, Gifu
  - Matsunami General Hospital, Gifu, Gifu
  - Hashima City Hospital, Hashima, Gifu
  - Ogaki Municipal Hospital, Ogaki-shi, Gifu
  - Gunma University Graduate School of Medicine, Maebashi, Gunma
  - Gunma Cancer Center, Otashi, Gunma
  - National Hospital Organization Fukuyama Medical Center, Fukuyama, Hiroshima
  - Chugoku Central Hospital of the Mutual Aid Association of Public School Teachers, Fukuyama, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Kure Medical Center, Kure, Hiroshima
  - Miyoshi Central Hospital, Miyoshi, Hiroshima
  - Asahikawa Medical College, Asahikawa, Hokkaido
  - Otaru Ekisaikai Hospital, Asahikawa, Hokkaido
  - Hakodate Goryoukaku Hospital, Hakodate, Hokkaido
  - Hirosaki University, School of Medicine, Otaru-shi, Hokkaido
  - Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - Sapporo Medical University, Sapporo, Hokkaido
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Hokkaido University Graduate School of Medicine, Sapporo, Hokkaido
  - Akashi Municipal Hospital, Akashi, Hyōgo
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Ako City Hospital, Akou, Hyōgo
  - Hyogo Prefectural Amagasaki Hospital, Amagasaki, Hyōgo
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Himeji St. Mary's Hospital, Himeji, Hyōgo
  - Himeji Central Hospital, Himeji, Hyōgo
  - Kinki Central Hospital, Itami, Hyōgo
  - Kakogawa Municipal Hospital, Kakogawa, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kobe City General Hospital, Kobe, Hyōgo
  - Shakai Hoken Kobe Central Hospital, Kobe, Hyōgo
  - Nishi-Kobe Medical Center, Kobe, Hyōgo
  - Kobe West City Hospital, Kobe, Hyōgo
  - Kobe Medical Center, Kobe, Hyōgo
  - Sano Hospital, Kobe, Hyōgo
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Hyogo Prefectural Awaji Hospital, Sumoto, Hyōgo
  - Takarazuka Municipal Hospital, Takarazuka, Hyōgo
  - Higashi Takarazuka Satoh Hospital, Takarazukai, Hyōgo
  - Public Shiso General Hospital, Yamsakicho, Hyōgo
  - National Hospital Organization Mito Medical Center, Ibaraki, Ibaraki
  - Mito Saiseikai General Hospital, Mito, Ibaraki
  - Tsuchiura Kyodo General Hospital, Tsuchiura, Ibaraki
  - Kanazawa Medical University, Kahoku-gun, Ishikawa-ken
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital, Morioka, Iwate
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Kagawa University Hospital, Hiragi, Kagawa-ken
  - Kagawa Rosai Hospital, Marugame, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Nanpuh Hospital, Kagoshima, Kagoshima-ken
  - Kanagawa Prefectural Ashigawa-kami Hospital, Ashigarakami-gun, Kanagawa
  - Chigasaki Municipal Hospital, Chigasaki, Kanagawa
  - Fujisawa City Hospital, Fujisawa-shi, Kanagawa
  - Kitasato University School of Medicine, Kanagawa, Kanagawa
  - Kanto Rosai Hospital, Kawasaki, Kanagawa
  - Nippon Medical School Musashikosugi Hospital, Kawasaki, Kanagawa
  - Saint Marianna University School of Medicine, Kawasaki, Kanagawa
  - Sagamihara National Hospital, Sagamihara, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Social Insurance Yokohama Central Hospital, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Saiseikai Yokohama City Nanbu Hospital, Yokohama, Kanagawa
  - Yokohama City Hospital, Yokohama, Kanagawa
  - St. Marianna University Yokohama City Seibu Hospital, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - International Goodwill Hospital, Yokohama, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - Kochi Health Sciences Center, Kochi, Kochi
  - Kochi Medical School, Nankoku, Kochi
  - Kumamoto University Faculty of Medical and Pharmaceutical Sciences, Kumamoto, Kumamoto
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - National Hospital Organization - Kumamotominami Hospital, Uki, Kumamoto
  - Japan Labor Health and Welfare Organization Kumamoto Rosai Hospital, Yashiro, Kumamoto
  - Yatsushiro Health Insurance General Hospital, Yatsushiro, Kumamoto
  - Kyoto First Red Cross Hospital, Higashiyama-ku, Kyoto
  - Kyoto Second Red Cross Hospital, Kanigyou-ku, Kyoto
  - Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Nishijin Hospital, Kyoto, Kyoto
  - National Hospital Organization - Kyoto Medical Center, Kyoto, Kyoto
  - Kyoto-Katsura Hospital, Kyoto, Kyoto
  - Nantan General Hospital, Nantan, Kyoto
  - Kyoto University Hospital, Sakyo-ku, Kyoto
  - Mie University Graduate School of Medicine, Thu-shi, Mie-ken
  - Miyagi Cancer Center, Natori-shi, Miyagi
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Tohoku University Graduate School of Medicine, Sendai, Miyagi
  - Tohoku Rosai Hospital, Sendai, Miyagi
  - Sendai Medical Center, Sendai, Miyagi
  - Iida Municipal Hospital, Iida, Nagano
  - Showa-Inan General Hospital, Komagane, Nagano
  - Aizawa Hospital, Matsumoto, Nagano
  - Nagano Municipal Hospital, Nagano, Nagano
  - Hokushin Hospital, Nakano, Nagano
  - Nagasaki University Hospital, Magasaki-shi, Nagasaki
  - Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki, Nagasaki
  - National Hospital Organization Nagasaki Medical Center, Ōmura, Nagasaki
  - Sasebo City General Hospital, Sasebo-shi, Nagasaki
  - Nara Medical University Cancer Center, Kashihara, Nara
  - Saiseikai Nara Hospital, Nara, Nara
  - Kenseikai Nara Coloproctology Center, Yamatotakada, Nara
  - Nagaoka Chuo General Hospital, Nagaoka, Niigata
  - Saiseikai Niigata Daini Hospital, Niigata, Niigata
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Oita University Hospital, Yufu-shi, Oita Prefecture
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kawasaki Medical School, Kurashiki-shi, Okayama-ken
  - Okayama University Medical School, Okayama, Okayama-ken
  - Nakagami Hospital, Okinawa, Okinawa
  - Hoshigaoka Koseinenkin Hospital, Hirakata, Osaka
  - Izumiotsu Municipal Hospital, Izumiōtsu, Osaka
  - Rinku General Medical Center, Izumisano, Osaka
  - Minoh City Hospital, Mino, Osaka
  - Kansai Medical University Takii Hospital, Moriguchi, Osaka
  - Kitano Hospital, Osaka, Osaka
  - Osaka City Juso Hospital, Osaka, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka Saiseikai Noe Hospital, Osaka, Osaka
  - Otemae Hospital, Osaka, Osaka
  - Osaka Police Hospital, Osaka, Osaka
  - Higashi Sumiyoshi Morimoto Hospital, Osaka, Osaka
  - Nissay Hospital, Osaka, Osaka
  - Osaka Kosei Nenkin Hospital, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Minamiosaka Hospital, Osaka, Osaka
  - Sakai Municipal Hospital, Sakai, Osaka
  - Bell Land General Hospital, Sakai, Osaka
  - Osaka Rosai Hospital, Sakai-shi, Osaka
  - Kinki University School of Medicine, Sayama, Osaka
  - Suita Municipal Hospital, Suita-shi, Osaka
  - Osaka Medical College, Takatsuki, Osaka
  - Saiseikai Tondabayashi Hospital, Tondabayashi, Osaka
  - Saga Prefectural Hospital Koseikan, Saga, Saga-ken
  - Fukaya Red Cross Hospital, Fukaya, Saitama
  - Hasuda Hospital, Hasuda, Saitama
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Saitama Medical School Hospital, Kawagoe-shi, Saitama
  - Kitasato Institute Medical Center Hospital, Kitamoto, Saitama
  - Saitama Social Insurance Hospital, Saitama, Saitama
  - Omiya Medical Center ofJichi Medical School, Saitamaken, Saitama
  - National Hospital Organization - Nishisaitama-Chuo National Hospital, Tokorozawa, Saitama
  - National Defense Medical College, Tokorozawa, Saitama
  - Otsu Municipal Hospital, Ōtsu, Shiga
  - Shiga University of Medical Science, Ōtsu, Shiga
  - Shimane Prefectural Central Hospital, Izumo-shi, Shimane
  - Fujieda Municipal General Hospital, Fujieda, Shizuoka
  - Hamamatsu University School of Medicine, Hamamatsu, Shizuoka
  - Shizuoka City Hospital, Shizuoka, Shizuoka
  - Shizuoka Municipal Shimizu Hospital, Shizuoka, Shizuoka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Yaizu Municipal Hospital, Yaizu, Shizuoka
  - Ohtawara Red Cross Hospital, Ohtawawa, Tochigi
  - Dokkyo University School of Medicine, Shimotsuga-gun, Tochigi
  - Jichi Medical School, Shimotsuke-shi, Tochigi
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Anan Kyoei Hospital, Anan, Tokushima
  - Tokushima University Hospital, Tokushima, Tokushima
  - Juntendo University School of Medicine, Bunkyo-ku, Tokyo
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - Tokyo Metropolitan Fuchu Hospital, Fuchū, Tokyo
  - Higashiyamato General Hospital, Higashiyamato, Tokyo
  - Tokyo-Kita Social Insurance Hospital, Kita-ku, Tokyo
  - Showa General Hospital, Kodaira, Tokyo
  - Daisan Hospital, Komae, Tokyo
  - Toho University Ohashi Hospital, Meguro-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - Kyorin University School of Medicine - Mitaka Campus, Mitaka, Tokyo
  - Nakano General Hospital, Nakano City, Tokyo
  - Social Insurance Chuo General Hospital, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University, Shinjyuku-ku, Tokyo
  - Mita Hospital at the International University of Health and Welfare, Tokyo, Tokyo
  - Tokyo Medical and Dental University, Tokyo, Tokyo
  - Nippon Medical School, Tokyo, Tokyo
  - Tokyo Metropolitan - Komagome Hospital, Tokyo, Tokyo
  - Tokyo Women's Medical University Medical Center East, Tokyo, Tokyo
  - Metropolitan Bokutoh Hospital, Tokyo, Tokyo
  - Showa University Toyosu Hospital, Tokyo, Tokyo
  - NTT Kanto Medical Center, Tokyo, Tokyo
  - Toho University School of Medicine, Tokyo, Tokyo
  - Japanese Red Cross Medical Center, Tokyo, Tokyo
  - National Hospital Organization - Tokyo Medical Center, Tokyo, Tokyo
  - International Medical Center of Japan, Tokyo, Tokyo
  - Teikyo University School of Medicine, Tokyo, Tokyo
  - Jikei University School of Medicine Hospital, Tokyo, Tokyo
  - Takasago Kyoritsu Hospital, Tokyo, Tokyo
  - Tottori University - Faculty of Medicine, Yonago, Tottori
  - Koseiren Takaoka Hospital, Takaoka-shi, Toyama
  - Toyama Red Cross Hospital, Toyama, Toyama
  - Toyama Prefectural Central Hospital, Toyama, Toyama
  - Shingu Municipal Medical Center, Shingū, Wakayama
  - Social Insurance Kinan Hospital, Tanabe, Wakayama
  - Japan Labor Health and Welfare Organization Wakayama Rosai Hospital, Wakayama, Wakayama
  - Wakayama Medical University, Wakayama, Wakayama
  - Yamagata Prefectural Central Hospital, Yamagata, Yamagata
  - Yamagata Saisei Hospital, Yamagata, Yamagata
  - Yamagata University Hospital, Yamagata, Yamagata
  - National Hospital Organization - Kanmon Medical Center, Shimonoseki, Yamaguchi
  - Shimonoseki Kosei Hospital, Shimonoseki, Yamaguchi
  - Yamaguchi University Graduate School of Medicine, Ube, Yamaguchi
  - University of Yamanashi Faculty of Medicine, Chu-o-shi, Yamanashi
  - Ageo Central General Hospital, Ageo
  - Saiseikai Hiroshima Hospital, Aki-Gun
  - Northern Fukushima Medical Center, Date
  - Chugoku Electric Power Hospital, Hiroshima
  - Hiroshima Red Cross Hospital and Atomic-bomb Survivors Hospital, Hiroshima
  - Hokkaido Chuo Rosai Hospital, Iwamizawa
  - Osaka Minami Medical Center, Kawachi-Nagano
  - Kiryu Kosei General Hospital, Kiryū
  - Kobe Ekisaikai Hospital, Kobe
  - Konan Kosei Hospital, Kōnan
  - Southern TOHOKU research Institute for Neuroscience, Kōriyama
  - Saiseikai Matsusaka General Hospital, Matsusaka
  - Muroran City General Hospital, Muroran
  - Kyoritsu General Hospital, Nagoya
  - Nakatsu Municipal Hospital, Nakatsu
  - Nara Prefectual Nara Hospital, Nara
  - Numazu City Hospital, Numazu, Shizuoka
  - Yodogawa Christian Hospital, Osaka
  - Osaka Red Cross Hospital, Osaka
  - NTT West Osaka Hospital, Osaka
  - Oita Red Cross Hospital, Ōita
  - Almeida Memorial Hospital, Ōita
  - Oita Prefectural Hospital, Ōita
  - Hakodate Municipal Hospital, Sendai
  - Miyagi Social Insurance Hospital, Sendai
  - Japanese Red Cross Sendai Hospital, Sendai
  - Kawakita General Hospital, Suginami-ku
  - Niigata Prefectural Tokamachi Hospital, Tōkamachi
  - Japanese Red Cross Society, Wakayama
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama
  - Yokohama City Minato Red Cross Hospital, Yokohama
  - Hitachi Yokohama Hospital, Yokohama

REFERENCES:
- [Derived] Ueno H, Ishiguro M, Nakatani E, Ishikawa T, Uetake H, Matsuda C, Nakamoto Y, Kotake M, Kurachi K, Egawa T, Yasumasa K, Murata K, Ikawa O, Shinji S, Murotani K, Matsui S, Teramukai S, Tomita N, Sugihara K; SACURA Study Group. Prospective Multicenter Study on the Prognostic and Predictive Impact of Tumor Budding in Stage II Colon Cancer: Results From the SACURA Trial. J Clin Oncol. 2019 Aug 1;37(22):1886-1894. doi: 10.1200/JCO.18.02059. Epub 2019 Jun 10. PMID 31180819
- [Derived] Matsuda C, Ishiguro M, Teramukai S, Kajiwara Y, Fujii S, Kinugasa Y, Nakamoto Y, Kotake M, Sakamoto Y, Kurachi K, Maeda A, Komori K, Tomita N, Shimada Y, Takahashi K, Kotake K, Watanabe M, Mochizuki H, Nakagawa Y, Sugihara K; SACURA Study Group. A randomised-controlled trial of 1-year adjuvant chemotherapy with oral tegafur-uracil versus surgery alone in stage II colon cancer: SACURA trial. Eur J Cancer. 2018 Jun;96:54-63. doi: 10.1016/j.ejca.2018.03.009. Epub 2018 Apr 17. PMID 29677641
- [Derived] Ishiguro M, Mochizuki H, Tomita N, Shimada Y, Takahashi K, Kotake K, Watanabe M, Kanemitsu Y, Ueno H, Ishikawa T, Uetake H, Matsui S, Teramukai S, Sugihara K. Study protocol of the SACURA trial: a randomized phase III trial of efficacy and safety of UFT as adjuvant chemotherapy for stage II colon cancer. BMC Cancer. 2012 Jul 7;12:281. doi: 10.1186/1471-2407-12-281. PMID 22769569